CLINICAL TRIAL: NCT02447796
Title: A Comparative Study of Dexmedetomidine and Propofol As Sole Sedative Agent for Patients With End-Stage Renal Disease Undergoing Arteriovenous Fistula Surgery
Brief Title: Dexmedetomidine and Propofol As Sole Sedative Agent for Patients Undergoing Arteriovenous Fistula Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Ozmete, Medical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA 15/60
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Arteriovenous Fistula
Keywords: (AVF); surgery
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): Propofol was administered at 1 mg/kg over a 10-min period followed by a continuous infusion at a rate of 1-1.5 mg/kg/h until the the begining of skin suture (n=24)
  Interventions: Drug: Propofol
- Dexmedetomidine (DEX) (Active Comparator): DEX was administered at 1 μg/kg over a 10-min period followed by a continuous infusion at a rate of 1-1.5 μg/kg/h until the begining of skin suture (n=24)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Propofol was administered at 1 mg/kg over a 10-min period followed by a continuous infusion at a rate of 1-1.5 mg/kg/h until the the begining of skin suture (n=24).
  Other Names: Pofol
  Arms: Propofol
Drug: Dexmedetomidine — DEX was administered at 1 μg/kg over a 10-min period followed by a continuous infusion at a rate of 1-1.5 μg/kg/h until the begining of skin suture (n=24).
  Other Names: Precedex
  Arms: Dexmedetomidine (DEX)

SUMMARY:
The investigators designed a prospective randomized study to compare the conventionally used sedative drug propofol with a latest alternative dexmedetomidine (DEX), in patients with end-stage renal disease undergoing arteriovenous fistula (AVF) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were patients undergoing arteriovenous fistula (AVF) surgery aged between 20-70 with end stage renal failure on dialysis treatment.

Exclusion Criteria:

* Exclusion criteria were decompensated respiratory or heart failure, liver failure, obesity (body mass index>30), severe obstructive sleep apnea, need for additional different drugs for sedation, chronic use of alcohol, opioids or other sedative drugs,mental disorders, cognitive disorders, language problems and history of allergy to any medications used in this study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse effects such as respiratory and hemodynamic events | up to 24 hours postoperative

SECONDARY OUTCOMES:
The sedation onset time with using BIS and recovery times during the procedure. | up to 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof md, Principal Investigator — Baskent University School of Medicine
Locations (1):
- Baskent University School of Medicine Adana Research and Teaching Center, Adana, Turkey (Türkiye)